CLINICAL TRIAL: NCT05339919
Title: The Effect of Sarcopenia on Hepatocellular Carcinoma After Hepatectomy
Brief Title: Relationship Between Liver Cancer and Sarcopenia
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Collaborators: Qilu Hospital of Shandong University (Other); The Second Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Gang Chen, MD, Clinical Professor, Principal Investigator, First Affiliated Hospital of Wenzhou Medical University
Other Study IDs: sarcopenia
Record Dates: First submitted 2022-04-09; First posted 2022-04-21 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Liver Cancer; Sarcopenia
Keywords: Sarcopenia; Liver cancer; Hepatectomy; Short-term outcomes; Long-term outcomes
MeSH Terms: conditions — Liver Neoplasms; Sarcopenia | interventions — Walking Speed

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — night soil；whole blood；Tissue specimen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: gait speed; ct scan;grip strength and chair stand test — The chair stand test was administered, and the time required for the patient to stand five times from a sitting position without using the arms was measured. CT scan was to scan the patient's third lumbar level. For the gait speed test, the time that patients spent walking 8 meters on a flat indoor floor at usual walking speed was measured.Grip strength test:the dominant hand and the nondominant hand were measured twice intermittently (kg), and the average value of 4 values was obtained.

SUMMARY:
By tracking the short-term and long-term results of patients after hepatectomy, the difference of short-term results between patients with sarcopenia and patients without sarcopenia was analyzed, and the correlation between sarcopenia and short-term and long-term results of patients after hepatectomy was explored, so as to improve people's awareness of sarcopenia and pay attention to its prevention and treatment.

DETAILED DESCRIPTION:
All implementation details are based on the newest EWGSOP definition. The investigators consecutively admitted patients the questionnaire and evaluated the assessment of muscle strength (grip strength test and chair stand test), muscle quantity (L3 plane total skeletal muscle area) and physical performance (gait test) following the F-A-C-S approach, to confirm patients with sarcopenia accurately. And by tracking the short-term and long-term outcomes of patients after hepatectomy, the differences were analyzed and the relationship between sarcopenia and liver cancer was explored.

ELIGIBILITY:
Inclusion Criteria:

* Patients with preoperative clinical diagnosis of liver cancer
* No cancer other than liver cancer has been diagnosed
* Age ≥18 years

Exclusion Criteria:

* Patients who could not complete the standard tests and questionnaires
* Patients who did not accept liver resection after evaluation of treatment plan
* Patients who had other concomitant preoperative causes of muscle weakness (injury, fracture, stroke, etc.)
* Patients who missing CT data or CT scan did not reach the level of the third lumbar vertebra (L3)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with preoperative clinical diagnosis of liver cancer admitted to the hepatobiliary surgery department and received standard tests and questionnaires.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-08-11 (Actual); Study Completion 2025-08-28 (Estimated)

PRIMARY OUTCOMES:
Short-term postoperative results | 3 months
  Postoperative complications；90 days readmission rate
Long-term results after operation | 10 years
  Overall survival; Disease free survival

SECONDARY OUTCOMES:
Postoperative hospitalization time | 2 months
  Time window from the day of operation to the day of discharge.
Hospitalization expenses | 2 months
  All hospitalization expenses, including drug expenses, operation expenses, anesthesia expenses, nursing expenses and other expenses.

CONTACTS AND LOCATIONS:
Overall Officials: Gang Chen, M.D., Principal Investigator — First Affiliated Hospital of Wenzhou Medical University
Locations (1):
- Gang Chen, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No